CLINICAL TRIAL: NCT03645018
Title: A Monocenter Prospective No-profit Interventional Study for Lung Cancer Early Diagnosis With Tomosynthesis: Re-evaluation of Lung Nodule Detection Rate at 5 Years
Brief Title: Lung Cancer Early Diagnosis With Digital Tomosynthesis: Re-evaluation of Lung Nodule Detection Rate at 5 Years
Acronym: SOS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Collaborators: Fondazione CRC - Cuneo (Unknown); University of Turin, Italy (Other)
Responsible Party: Principal Investigator, MAURIZIO GROSSO, Head of Radiology Dept., Ospedale Santa Croce-Carle Cuneo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOS2
Record Dates: First submitted 2018-07-20; First posted 2018-08-24 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Lung Cancer
Keywords: lung; cancer; early diagnosis; DTS
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Disease | interventions — Diagnosis

STUDY DESIGN:
Intervention Model Description: Monocenter prospective no-profit single group interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnosis with tomosynthesis (DTS) (Experimental): Single arm.
  Population: Subjects enrolled in previously closed SOS trial (high risk subjects for lung cancer) without confirmed lung cancer.
  Interventions: Diagnostic Test: diagnosis with tomosynthesis

INTERVENTIONS:
Diagnostic Test: diagnosis with tomosynthesis — Re-evaluation of lung nodule detection rate at 5 years in patients with early diagnosis of lung cancer

SUMMARY:
Lung cancer is the leading cause of cancer-related death around the world, it represents 13% of all new cancer diagnoses. The lung cancer incidence is gradually increasing, especially among women and young people, but the fraction of cured patient remains low. In 80% of cases lung cancer, in early phase, is treatable only with surgery without chemotherapy or adjuvant radiotherapy and the survival perspective at five years exceeds 70%. Several scientific guidelines recommends chest CT (computed tomography) in lung cancer screening. Digital tomosynthesis (DTS) is a limited angle tomography that allows reconstruction of coronal images from a set of projection acquired over a small angle of X-ray tube movement. Several studies demonstrates that DTS is a reasonable alternative to the CT and allows a better evaluation of suspects nodules compared to conventional chest RX.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death around the world. In 2008 there were nearly 1.6 million new cases worldwide, accounting for the 12.7% of all new cancer diagnoses. Despite decreasing trends in smoking and resulting decrease in lung cancer mortality, the population at risk for lung cancer continues to be large. In the past years several programs have been developed to screen for lung cancer using low-dose chest computed radiography (CT). However, only recently different studies demonstrated a clear reduction in mortality. In particular, NLST low dose CT screening trial demonstrated a 6.7% reduction in the death rate compared to chest X-ray with a positive screening test rate for lung cancer detection of 24.2%, compared to 6.9% for conventional X-ray. Digital tomosynthesis (DTS) is a limited angle tomography that allows reconstruction of multiple image planes from a set of projection data acquired over a relatively small angle of X-ray tube movement. Although it does not have the spatial depth resolution of computed tomography, it provides high-resolution images in the sagittal planes at a lower dose and cost than CT. Several studies have shown that DTS offers advantages over conventional chest X-ray and comparable of those of CT. The Studio OSservazionale (SOS) was a clinical trial conducted within Santa Croce e Carle Hospital analysing smokers and former smokers aged 45-80 with no cancer diagnosis. All the subjects in whom a suspicious nodule was detected by DTS underwent diagnostic CT. The SOS study demonstrated that baseline DTS detected pulmonary abnormalities in 14.5% and lung cancer in 1.0% of the subjects, comparable to results that are obtained in CT screening programs. A second DTS, within the same study, executed one year later reported pulmonary abnormalities in 0.7% and lung cancer in 0.3% of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* current or former smoker status;
* for former smokers, the maximum time since quitting smoking must be below 10 years;
* smoking history of at least 20 pack-years;
* age 45-80 years;
* no previous history of cancer in the 10 years before the beginning of the study;
* be able to stand and hold the breath for 11 seconds during image acquisition;
* previous participation to SOS trial.

Exclusion Criteria:

* pregnancy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1341 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the lung cancer detection rate in the population of high risks subjects previously enrolled in lung cancer screening trial with chest digital tomosynthesis (SOS trial). | 1 year
  Lung cancer detection rate (primary endpoint)

SECONDARY OUTCOMES:
Percentage of lung cancer addressed to radical surgery treatment | 1 year
Sensitivity of DTS evaluating the number of lung cancer occurred in the population of SOS study in the last 5 years | 1 year
Mortality | 1 year
OS | 1 year
  Overall survival
QoL: quality of life: Percentage of partecipants changing their smoking habits | 1 year
  Percentage of partecipants changing their smoking habits after trial

CONTACTS AND LOCATIONS:
Locations (1):
- OSCroceCarle, Cuneo, CN, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Terzi A, Bertolaccini L, Viti A, Comello L, Ghirardo D, Priotto R, Grosso M; SOS Study Group. Lung cancer detection with digital chest tomosynthesis: baseline results from the observational study SOS. J Thorac Oncol. 2013 Jun;8(6):685-92. doi: 10.1097/JTO.0b013e318292bdef. PMID 23612466
- [Result] Bertolaccini L, Viti A, Tavella C, Priotto R, Ghirardo D, Grosso M, Terzi A; SOS Study Group. Lung cancer detection with digital chest tomosynthesis: first round results from the SOS observational study. Ann Transl Med. 2015 Apr;3(5):67. doi: 10.3978/j.issn.2305-5839.2015.03.41. PMID 25992366

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT03645018/Prot_SAP_002.pdf